CLINICAL TRIAL: NCT02857920
Title: Combination of Bevacizumab and Allogeneic NK Immunotherapy for Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-Bevacizumab
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2018-08

CONDITIONS: Malignant Solid Tumour
Keywords: Vascular Endothelial Growth Factor (VEGF) antibody; solid tumor; NK Immunotherapy
MeSH Terms: interventions — Bevacizumab

ARMS (2):
- Bevacizumab and NK immunotherapy (Experimental): In this group, the patients will receive regular Bevacizumab treatment in combination with multiple NK immunotherapies. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Bevacizumab; Biological: NK immunotherapy
- Bevacizumab (Active Comparator): In this group, the patients will receive regular Bevacizumab treatment to control the tumor growth. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 7.5 mg/kg, i.v, once every 3 weeks (continuous)
  Other Names: Anti-VEGF, Avastin
Biological: NK immunotherapy — Each treatment: 8~10 billion cells in all, transfusion in 3 times, i.v.
  Arms: Bevacizumab and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of Bevacizumab plus allogeneic natural killer (NK) immunotherapy to many kinds of recurrent solid tumors.

DETAILED DESCRIPTION:
By enrolling patients with recurrent solid tumors adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using Bevacizumab and NK cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
PFS | 1 year
  PFS was defined as the interval between treatment initiation and local relapse
OS | 3 years
  OS was calculated as the interval from treatment initiation to death.

SECONDARY OUTCOMES:
Tumor size | 3 months
  The tumor responses of the enrolled patients were assessed by CT in accordance with RECIST v1.1.Institute Common Terminology Criteria for Adverse Events (v4.0).
CTC | 3 months
  The absolute number of CD45-CK+ CD326+ cells was used to quantitate the CTC levels.
PD-1 | 3 months
  Peripheral blood (6 mL) was obtained from healthy donors and patients before treatment and 90 days after treatment for the detection of PD-1

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Fuda cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China